CLINICAL TRIAL: NCT07056127
Title: Antimicrobial Impact of Various Root Canal Final Irrigation Activation Techniques (Clinical Study)
Brief Title: Antimicrobial Impact of Various RC Final Irrigation Activation Techniques
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Randa Ahmed Abdo Elsobky, Assistant teacher, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Irrigant activaion
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Root Canal Final Irrigation Activation Techniques
Keywords: Irrigant activation, ultrasonic, xp-endo finisher
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- manual dynamic agitation (Active Comparator)
  Interventions: Other: manual dynamic agitaion
- ultrasonic activation (Active Comparator)
  Interventions: Other: ultrasonic activation
- xp-endo finisher (Active Comparator)
  Interventions: Other: xp-endo finisher
- laser (Active Comparator)
  Interventions: Other: laser

INTERVENTIONS:
Other: manual dynamic agitaion — 5 mL of 2.5% NaOCl solution will be activated with a well-fitting gutta-percha cone that will be placed to full working length and then will be moved in push-pull strokes of 2 mm amplitude at a frequency of 100 strokes in about 1 min
  Arms: manual dynamic agitation
Other: ultrasonic activation — 5 mL of 5.25% NaOCl solution will be activated with PUI using a #20 endosonic ﬁle that will be driven by an ultrasonic device on medium power setting for 1 minute and inserted 1 mm short of the working length
  Arms: ultrasonic activation
Other: xp-endo finisher — 5 mL of 5.25% NaOCl solution will be activated with XP-Endo Finisher which will be used in the canal for 1 minute at 800 rpm and 1 Ncm up to the working length and in slow up-and-down movements at 7-8mm length according to the manufacturer's recommendations
  Arms: xp-endo finisher
Other: laser — First, root canals will be filled with 0.5 mL of 0.05% ICG dye and left in place for 1 minute as preirradiation time. A #20 laser fiber will be inserted into the root canals to the working length. Then infrared diode laser with a wave length of 810 nm will be used to activate the dye for 30 seconds. For activation, circular movements will be performed along with the fiber removal movement . After the first activation, dye will be reintroduced, the laser fiber will be inserted again, and a new activation cycle of 30 seconds will be performed similarly to the previous one
  Arms: laser

SUMMARY:
This randomized clinical study aims to evaluate microbial reduction in root canals after using different final irrigation activation techniques including passive ultrasonic irrigation, XP-endo Finisher file and Laser ablation with Indocyanine green dye in comparison to manual dynamic activation.

ELIGIBILITY:
Inclusion Criteria:

• Vital/non vital single rooted teeth with single root canal with nearly the same apical diameter requiring root canal treatment.

* Teeth with sound periodontal apparatus.

Exclusion Criteria:

* • Teeth with anatomic anomilies.

  * Retreatment cases
  * Pregnant patients

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
bacterial count | 24-48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No